CLINICAL TRIAL: NCT00428506
Title: Albumin 4 gr/L vs 8 gr/L in the Prevention of Post-Paracentesis Circulatory Dysfunction in Cirrhotic Patients With Ascites
Brief Title: Albumin 4 gr/L vs 8 gr/L in the Prevention of Post-Paracentesis Circulatory Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: University of Turin, Mario Rizzetto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALB-PPCD
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Tense Ascites in Cirrhosis
Keywords: ascites; cirrhosis; post-paracentesis circulatory dysfunction; albumin; portal-hypertension
MeSH Terms: conditions — Ascites; Fibrosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: albumin 4 gr/L ascites removed — albumin 4 gr/L ascites removed
Drug: albumin 8 gr/L ascites removed — albumin 8 gr/L ascites removed

SUMMARY:
The purpose of this study is to determine whether the infusion of albumin 4 gr per liter of ascites removed is as effective as the infusion of albumin 8 gr per liter of ascites removed in the prevention of post-paracentesis circulatory dysfunction

DETAILED DESCRIPTION:
Large-volume paracentesis associated with plasma volume expansion is the first-line treatment of tense ascites in cirrhotic patients. When paracentesis is performed without volume expansion, an high proportion of patients develop a complication named post-paracentesis circulatory dysfunction, which is characterized by a marked activation of the renin-angiotensin-aldosterone system. PPCD has been associated with renal impairment, rapid recurrence of ascites and shorter survival. Infusion of albumin is very effective in the prevention of PPCD, but has sever inherent drawbacks: the theoretical possibility of transmission of infectious diseases and the high costs. Other synthetic plasma volume expanders have been proposed in the last decades, but they are less effective than albumin when large (> 5 L) volume paracentesis are performed. Albumin is conventionally given in a dosage of 8 gr per liter of ascites removed; however no information has yet been reported on the use of lower dosages of albumin in this context. This would be interesting, because of the obvious advantages in terms of costs reduction.

The aim of the present study is to compare the efficacy of the infusion of albumin 4 gr vs 8 gr per liter of ascites removed in the prevention of PPCD.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis and ascites submitted to paracentesis > 5 liters
* Age: 18-75 years
* Informed written consent

Exclusion Criteria:

* Multinodular HCC (> 3 nodules)
* Portal vein thrombosis
* Ongoing bacterial infection
* Ongoing or recent (less than one week) bleeding
* Cardio-pulmonary failure
* Hepatorenal syndrome type 1
* Severe coagulopathy: platelets < 30.000/mm3 and/or PT < 30%
* Ongoing treatment with vasoactive drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
renin-angiotensin-aldosterone activation | 4-6 days

SECONDARY OUTCOMES:
renal function | 4-6 days

CONTACTS AND LOCATIONS:
Overall Officials: Mario Rizzetto, MD, Study Director — Division of Gastroenterology and Hepatology, San Giovanni Battista Hospital, Turin, Italy
Locations (1):
- San Giovanni Battista Hospital, Turin, Italy

REFERENCES:
- [Background] Sola-Vera J, Minana J, Ricart E, Planella M, Gonzalez B, Torras X, Rodriguez J, Such J, Pascual S, Soriano G, Perez-Mateo M, Guarner C. Randomized trial comparing albumin and saline in the prevention of paracentesis-induced circulatory dysfunction in cirrhotic patients with ascites. Hepatology. 2003 May;37(5):1147-53. doi: 10.1053/jhep.2003.50169. PMID 12717396
- [Background] Gines A, Fernandez-Esparrach G, Monescillo A, Vila C, Domenech E, Abecasis R, Angeli P, Ruiz-Del-Arbol L, Planas R, Sola R, Gines P, Terg R, Inglada L, Vaque P, Salerno F, Vargas V, Clemente G, Quer JC, Jimenez W, Arroyo V, Rodes J. Randomized trial comparing albumin, dextran 70, and polygeline in cirrhotic patients with ascites treated by paracentesis. Gastroenterology. 1996 Oct;111(4):1002-10. doi: 10.1016/s0016-5085(96)70068-9. PMID 8831595
- [Derived] Alessandria C, Elia C, Mezzabotta L, Risso A, Andrealli A, Spandre M, Morgando A, Marzano A, Rizzetto M. Prevention of paracentesis-induced circulatory dysfunction in cirrhosis: standard vs half albumin doses. A prospective, randomized, unblinded pilot study. Dig Liver Dis. 2011 Nov;43(11):881-6. doi: 10.1016/j.dld.2011.06.001. Epub 2011 Jul 8. PMID 21741331